CLINICAL TRIAL: NCT05558696
Title: A Phase 2 Multi-Center, Open Label Study to Assess the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Bomedemstat in Patients With Polycythemia Vera (PV)
Brief Title: A Study of Bomedemstat (MK-3543) in Participants With Polycythemia Vera (MK-3543-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3543-004; MK-3543-004 (Other: MSD); IMG-7289 (Other: Imagobio ID)
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Polycythemia Vera
Keywords: polycythemia vera; bomedemstat
MeSH Terms: conditions — Polycythemia Vera | interventions — bomedemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bomedemstat (Experimental): Participants will receive bomedemstat daily for 36 weeks and may qualify for additional treatment through Week 52 if deriving clinical benefit.
  Interventions: Drug: Bomedemstat

INTERVENTIONS:
Drug: Bomedemstat — Oral tablet
  Other Names: MK-3543; IMG-7289

SUMMARY:
This study will evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics of the orally administered lysine-specific demethylase 1 (LSD1) inhibitor bomedemstat, in participants with polycythemia vera (PV). At Week 36 of dosing, participants will be assessed for eligibility to receive additional treatment through Week 52. Participants deriving clinical benefit and safely tolerating bomedemstat will qualify for continued treatment at the Investigator's discretion.

DETAILED DESCRIPTION:
With Amendment 3, after all ongoing participants have reached 52 weeks of treatment, eligible participants may transition to a bomedemstat extension study if available. With Amendment 4, all secondary PK and patient reported outcome measures were designated as exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of Polycythemia Vera per World Health Organization (WHO) diagnostic criteria for myeloproliferative neoplasms
* Has a bone marrow fibrosis score of Grade 0 or Grade 1
* Has failed at least one standard cytoreductive therapy to lower hematocrit
* Has a life expectancy >36 weeks
* Has discontinued prior cytoreductive therapy for 2 weeks (4 weeks for interferon) prior to study drug initiation

Exclusion Criteria:

* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 3 or greater
* Has unresolved treatment related toxicities from prior therapies (unless resolved to ≤ Grade 1)
* Has an uncontrolled active infection
* Has a known human immunodeficiency virus (HIV) infection or active Hepatitis B or Hepatitis C virus infection
* Has evidence of increased risk of bleeding, including known bleeding disorders
* Is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to ~56 weeks
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with one or more AEs will be reported.
Number of participants who discontinued study intervention due to AEs | Up to ~52 weeks
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to AEs will be reported.
Number of participants with sustained change from baseline of hematocrit to <45% without concomitant phlebotomy at Week 36 | Baseline through Week 36
  Hematocrit will be analyzed by taking blood samples from participants at designated time points during the study. The number of participants who have achieved a sustained change from baseline of hematocrit to <45% without concomitant phlebotomy at Week 36 will be reported.

SECONDARY OUTCOMES:
Duration of reduction of hematocrit to <45% without phlebotomy | Baseline through Week 36
  Hematocrit will be analyzed by taking blood samples from participants at designated time points during the study. The duration of a reduction in hematocrit to <45% without phlebotomy up to Week 36 will be reported.
Number of participants with platelet count ≤ 450 x 10^9/L at Week 36 | Baseline through Week 36
  Platelet count will be analyzed by taking blood samples from participants at designated time points during the study. The percentage of participants who have a platelet count ≤450 X 10^9/L will be reported.
Duration of platelet count ≤ 450 x 10^9/L in participants at Week 36 | Baseline through Week 36
  Platelet count will be analyzed by taking blood samples from participants at designated time points during the study. The duration of the reduction of platelet count of ≤450 X 10^9/L in participants will be reported.
Number of participants with white blood cell (WBC) count of <10 x 10^9/L at Week 36 | Baseline through Week 36
  WBC count will be analyzed by taking blood samples from participants at designated time points during the study. The percentage of participants who have a WBC count of <10 X 10^9/L will be reported.
Duration of white blood cell (WBC) count <10 x 10^9/L in participants at Week 36 | Baseline through Week 36
  WBC count will be analyzed by taking blood samples from participants at designated time points during the study. The duration of the reduction of WBC count <10 X 10^9/L in participants will be reported.
Number of participants with thrombotic events | Baseline through Week 36
  Thrombotic events are defined as: new or recurrent acute myocardial infarction; unstable angina; stroke; transient ischemic attack (TIA); deep venous thrombosis (DVT); pulmonary embolism (PE); thrombotic digital ischemia; other thrombotic events such as peripheral limb ischemia or Budd-Chiari syndrome that are assessed to be due to underlying PV; other vascular occlusive events such as symptoms of cardiac, abdominal or peripheral limb ischemia supported by objective evidence of vessel disease and/or ischemia. The number of participants with thrombotic events will be reported.
Number of participants with major hemorrhagic events | Baseline through Week 36
  Hemorrhagic events are defined as: Major Bleeding (MB) Events such as fatal bleeding, and/or symptomatic bleeding in a critical area or organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in hemoglobin level of 2 g/dL or more, or leading to transfusion of 2 or more units of whole blood or red cells; Clinically Relevant Non-Major Bleeding (CRNMB) Events Leading to hospitalization or increased level of care or clinically important, prompting a face-to-face medical evaluation. The number of participants with hemorrhagic events will be reported.
Number of participants with a reduction in splenic volume in patients with an enlarged spleen at baseline | Baseline through Week 36
  Spleen volume will be measured by magnetic resonance imaging (MRI) (or computerized tomography [CT] if participant is not a candidate for MRI) of the abdomen according to standard procedures. The number of participants with a reduction in spleen volume by Week 36 will be reported.
Number of participants with progressive disease (PD) | Baseline through Week 36
  PD is defined as the worsening of PV to post-polycythemia vera myelofibrosis, myelodysplastic syndrome or transformation to acute myeloid leukemia. The number of participants with PD will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- United States (8):
  - BRCR Global ( Site 0120), Plantation, Florida
  - Hematology Oncology of the North Shore ( Site 0104), Skokie, Illinois
  - University of Michigan Comprehensive Cancer Center ( Site 0008), Ann Arbor, Michigan
  - Comprehensive Cancer Centers of Nevada - Peak ( Site 0118), Las Vegas, Nevada
  - Duke University Medical Center ( Site 0016), Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center ( Site 0103), Columbus, Ohio
  - OHSU Knight Cardiovascular Institute Cardiology Clinic - South Waterfront ( Site 0102), Portland, Oregon
  - Huntsman Cancer Hospital at the University of Utah ( Site 0119), Salt Lake City, Utah
- Australia (3):
  - Sunshine Coast Hematology and Oncology Clinic (Site 0506), Sunshine Coast, Queensland
  - Monash Medical Centre ( Site 0006), Clayton, Victoria
  - Royal Perth Hospital ( Site 0504), Perth, Western Australia
- United Kingdom (6):
  - Gloucestershire Royal Hospital ( Site 0205), Gloucester, England
  - United Lincolnshire Hospitals NHS Trust ( Site 0204), Lincoln, Great Britain
  - Imperial College London ( Site 0025), London, Great Britain
  - Boston Pilgrim Hospital ( Site 0207), Boston, Lincolnshire
  - Guys and St Thomas NHS Foundation Trust - Guys Hospital ( Site 0020), London, London, City of
  - Royal Gwent Hospital ( Site 0201), Newport, Wales

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26326&tenant=MT_MSD_9011